CLINICAL TRIAL: NCT06073145
Title: Non-invasive Monitoring of Blood Flow in the Brain by Using a Wearable Ultrasound Patch
Brief Title: Transcranial Doppler Using Wearable Ultrasound Patch
Acronym: TCD
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheng Xu, Associate Professor, University of California, San Diego
Other Study IDs: 805201
Record Dates: First submitted 2023-09-13; First posted 2023-10-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Medical Device Complication; Brain Injuries; Brain Diseases; Stroke; Vasospasm
MeSH Terms: conditions — Brain Injuries; Brain Diseases; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood flow monitoring in the brain: A group/cohort of 60 participants will be recruited. The group/cohort has a broad range distribution of different physiological parameters, such as age, gender, race, BMI, and etc.
  Interventions: Device: conventional transcranial Doppler probe and wearable ultrasound patch.

INTERVENTIONS:
Device: conventional transcranial Doppler probe and wearable ultrasound patch. — Comparison of the measurements from conventional transcranial Doppler probe and wearable ultrasound patch.

SUMMARY:
The main objective of this research is to measure the Doppler signal by the ultrasonic patch. Blood flow measurement is critical for vasospasm, stroke, and embolism monitoring on patients in the ICU or understanding the neurovascular coupling on different subjects. Currently, A conventional transcranial Doppler (TCD) probe is widely used for these applications. A headset design must be applied and fixed on the participants to obtain stable blood flow spectra. However, the TCD headset is operator dependent. The operator needs to be a trained expert and hold the ultrasound probe to get accurate blood flow velocity information. The stretchable and wearable non-invasive ultrasonic patch can not only free the operator's hands but can also provide long-term continuous monitoring, which is not possible by using the current operator-dependent ultrasound machine. The device can be conformal to the skin and attached to the skin surface.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* In relatively good health with no serious medical conditions.

Exclusion Criteria:

* Inability to sign the informed consent.
* History of the following conditions: Heart attack, low blood pressure, aortic stenosis/carotid artery stenosis (also known as heart valve disease), glaucoma (a group of eye conditions that damage the optic nerve) or retinopathy (a disease of the eye retina).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants without any serious medical conditions.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Device comparison to standard monitoring (conventional transcranial Doppler) | 1.5 years
  Clinical feasibility of the measurements from the non-invasive ultrasound patch in comparison to a conventional transcranial Doppler probe on 60 participants. Specifically, the blood flow specturm of different arterial segments including middle cerebral artery, anterior cerebral artery, posterior cerebral artery, vertebral artery, basal artery, internal carotid artery, and ophthalmic artery will be measured by the wearable ultrasound patch and the conventional transcranial Doppler probe. The agreement of these two device on peak systolic velocity, mean flow velocity, and end diastolic velocity of the measurements will be evaulated using the Bland-Altman plot.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Xu, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Structural and Materials Engineering (SME) building Room 310, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, and clinical study report will be shared and discussed in the research articles.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1.5 years
Access Criteria: Anyone can access it through research articles.